CLINICAL TRIAL: NCT07394608
Title: Use of Paired Non-Invasive Vagus Nerve Stimulation in Rehabilitation of Adolescents With Cerebral Palsy: An Open Label Safety Feasibility Trial
Brief Title: Paired Non-invasive VNS in Adolescent Cerebral Palsy Rehabilitation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, David Putrino, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY-25-01164
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-11

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Non-invasive VNS (Experimental): Non-invasive, transauricular, vagus nerve stimulation device will be used during physical therapy rehabilitation sessions
  Interventions: Device: Non-invasive taVNS

INTERVENTIONS:
Device: Non-invasive taVNS — Device activates the vagus through the ear. The device is controlled via the Vagustim mobile app, which connects using Bluetooth Low Energy (BLE).
  Other Names: Non-invasive, transauricular, vagus nerve stimulation device; Vagustim

SUMMARY:
This is an open-label safety and feasibility trial evaluating the use of paired non-invasive vagus nerve stimulation (VNS) and upper extremity (UE) rehabilitation in the motor impairment reduction of adolescent patients with spastic cerebral palsy.

ELIGIBILITY:
Inclusion criteria:

* Age 12-17 years old
* Diagnosis of spastic cerebral palsy
* Gross Motor Function Classification System (GMFCS) Level II-III (will be evaluated at screening)
* Jebsen Taylor Hand Function Test Score of <37.08 on the affected side at time of screening visit (will be evaluated at screening)
* Ability to communicate and follow two step commands at the time of screening
* Ability to provide assent as detailed in consent form and based on assessment using the University of California, San Diego Brief Assessment of Capacity to Consent

Exclusion criteria:

* Previous vagus nerve injury
* Less than 12 years old or greater than 18 years old
* History of left or bilateral vagotomy
* Current use of other implanted stimulation devices including but not limited to pacemaker, deep brain stimulator, implanted vagus nerve stimulators, cochlear implants, implantable cardiac defibrillators (ICDs)etc.
* Current use of any investigational devices or investigational drugs not otherwise specified - Past Medical History for any of the following:

  * Acute suicidal thinking or behavior
  * History of schizophrenia, schizoaffective disorder, or delusional disorders
  * History of rapid cycling bipolar disorder
  * Progressive neurological diseases
  * Cardiac arrhythmias or other abnormalities
  * History of dysautonomia including but not limited to orthostatic hypotension, postural orthostatic tachycardia syndrome, vasovagal syncope etc.
* GMFCS score of less than II or greater than III (will be evaluated at screening)
* Jebsen Taylor Hand Function Test Score of >37.08 on the affected side at time of screening visit (will be evaluated at screening)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of adverse event and serious adverse events | 12 months
  Safety is assessed by adverse event.

SECONDARY OUTCOMES:
Number of therapy sessions complete | end of therapy visits at Day 46
  Number of therapy sessions complete
Active training time per session | end of therapy visits at Day 46
  Number of minutes of training per session
Number of movement repetitions completed per session | end of therapy visits at Day 46
  Number of movement repetitions completed per session.
Jebsen Taylor Hand Function Test (JTHFT) | baseline Day 1, start of therapy Day 3, end of therapy Day 46, and 3, 6, 9, and 12 months
  The Jebsen Taylor Hand Function Test (JTHFT) is a standardized and objective measure of fine and gross motor hand functions that uses simulated activities of daily living (ADLs) assessed by time to completion; typically up to several minutes depending on impairment
BOT-2 | baseline Day 1, start of therapy Day 3, end of therapy Day 46, and 3, 6, 9, and 12 months
  The BOT-2 is a standardized assessment of motor proficiency in children and adolescents. It evaluates fine motor skills, manual dexterity, coordination, and motor integration through structured performance tasks.
  Fine Motor Precision (Upper Extremity) scored 0-41, higher score indicates better precision Fine Motor Integration (Upper Extremity) scored 0-45, higher score indicates better integration Manual Dexterity (Upper Extremity) scored 0- 45, higher score indicates better manual dexterity.
  Upper-Limb Coordination scored 0-30, higher score indicates better upper-limb coordination.
ABILHANDS | baseline Day 1, start of therapy Day 3, end of therapy Day 46, and 3, 6, 9, and 12 months
  ABILHAND is a patient-reported outcome measure that evaluates a person's perceived manual ability to perform daily bimanual activities. It assesses how difficult activities are to perform using both hands.
  The ABILHAND-Kids logit score ranges from -6 logits to +6 logits, higher score indicates better bimanual manual ability (tasks are perceived as easier).
Pediatric Evaluation of Disability (PEDI) | at 12 months
  The PEDI assesses functional abilities and performance in children across three domains: self-care, mobility, and social function. It measures both capability and caregiver assistance.
  Subscale range and full range uses scaled scores standardized to a 0-100 metric. Higher scores indicate better functional abilities and greater independence.
Pediatric Quality of Life Inventory (PedsQL) | baseline Day 1, start of therapy Day 3, end of therapy Day 46, and 3, 6, 9, and 12 months
  The PedsQL is a standardized patient-reported outcome measure assessing health-related quality of life in children across domains including physical, emotional, social, and school functioning.
  Subscales range and full scale scores are transformed to a 0-100 scale. Higher scores indicate better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: David Putrino, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- The Charles Lazarus Children's Abilities Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No: There is not a plan to make IPD available.